CLINICAL TRIAL: NCT04732728
Title: LUX-Dx Insertable Cardiac Monitor Remote Programming and Performance Study
Acronym: LUX-Dx PERFORM
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 92557593
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation; Syncope; Cryptogenic Stroke
MeSH Terms: conditions — Atrial Fibrillation; Syncope; Ischemic Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LUX-Dx PERFORM Study Enrollment: The first 227 subjects enrolled in the study belong to the "Safety Cohort". The number of subjects is required to fulfill the sample size requirement of the primary safety endpoint. The "Safety Cohort" subjects are not required to participate in the Holter study. Once the "Safety Cohort" enrollment is completed, all subsequent subjects are required to participate in the Holter study. All subjects who participate in the Holter study belong to the "Holter Cohort".

SUMMARY:
The LUX-Dx PERFORM Study had two primary objects which were (1) to characterize, in a general patient population, the utilization of the remote programming feature of the Boston Scientific (BSC) Insertable Cardiac Monitor (ICM) device and (2) to collect data to characterize the performance of arrhythmia detection algorithms. Data was also collected to characterize the ICM system related safety events.

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated to be implanted with the LUX-Dx ICM for one of the following reasons (grouped in three "Reason for Monitoring" subgroups): 1) Cryptogenic stroke, 2) Syncope, 3) AF management, Post-AF ablation, or Suspected AF
* Patient is willing to enroll and be monitored in LATITUDE Clarity.
* Patient is willing and able to be followed remotely via the ICM patient mobile app.
* Patient is willing and capable of providing informed consent (which is not to include the use of a legally authorized representative (LAR) for documentation of informed consent) and agrees to participate in all protocol required activities.
* Patient is age 18 years or above, or of legal age to give informed consent specific to state and national law.

The following inclusion criterion is applicable for patients participating in the Holter study:

• Patient can tolerate the adhesive used in the Holter monitoring for an extended period of time.

Exclusion Criteria:

* Patient is indicated for implantation of, or is currently implanted with an active implantable cardiac device (e.g., LVAD, ICD, CRT D, PPM*).
* Patient cannot tolerate a subcutaneous, chronically-inserted device due to medical condition.
* Patient has a documented life expectancy of less than 12 months (per investigator's discretion).
* Patient is known to be pregnant at the time of study enrollment (method of assessment upon investigator's discretion).
* Patient is currently enrolled in another clinical study including observational studies/registries, unless prior written approval from BSC is obtained. Mandatory governmental registries are accepted for co-enrollment without approval by BSC.

The following exclusion criteria are applicable for patients participating in the Holter study:

* Patient has known allergies to the adhesive materials or hydrogel used in the extended Holter monitoring.
* Patient has broken, damaged, or irritated skin over the chest area where the extended Holter monitor will be attached.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that have a known heart condition and are at risk of developing an abnormal heart rhythm, or have symptoms that may suggest a cardiac arrhythmia such as dizziness, palpitations, syncope, chest pain, and/or shortness of breath.
Sampling Method: Non-Probability Sample
Enrollment: 727 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Northern Arizona Healthcare, Flagstaff, Arizona
  - Arrythmia Research Group, Jonesboro, Arkansas
  - Scripps Memorial Hospital, La Jolla, California
  - Cardiology Associates Medical Group, Ventura, California
  - Cardiac Arrhythmia Service, Boca Raton, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - St. Luke's Idaho Cardiology Associates, Boise, Idaho
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Kansas City Arrhythmia Research LLC, Kansas City, Missouri
  - Cox Health, Springfield, Missouri
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Mount Sinai Morningside, New York, New York
  - North Carolina Heart and Vascular Research, Raleigh, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Presbyterian University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Monument Health Rapid City Hospital, Rapid City, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - PeaceHealth Southwest Medical, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LUX-Dx PERFORM Study Enrollment: The first 227 subjects enrolled in the study belonged to the "Safety Cohort". The number of subjects was required to fulfill the sample size requirement of the primary safety endpoint. The "Safety Cohort" subjects were not required to participate in the Holter study. Once the "Safety Cohort" enrollment was completed, all subsequent subjects were required to participate in the Holter study. All subjects who participated in the Holter study belong to the "Holter Cohort".
Period: Overall Study
Arm/Group | LUX-Dx PERFORM Study Enrollment
Started | 727
Completed | 579
Not Completed | 148
Not completed — Death | 12
Not completed — Withdrawn | 136

BASELINE CHARACTERISTICS:
Arm/Group | LUX-Dx PERFORM Study Enrollment
Number analyzed (Participants) | 727
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 372
  Male | 355
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Categories are not mutually exclusive.
  Participants
    White | 634
    Black or African American | 60
    Asian | 5
    American Indian or Alaska Native | 1
    Native Hawaiian or other Pacific Islander | 1
    Race - Other | 2
    Not disclosed | 27
    Ethnicity Hispanic or Latino - Mexican | 15
    Ethnicity Hispanic or Latino - Puerto Rican | 1
    Ethnicity Hispanic or Latino - Other | 11

OUTCOME MEASURES:

1. Primary Outcome: ICM System-related Complication-free Rate at 30 Days Post-implant
Time Frame: 30 days
Population: The acute primary safety endpoint was the LUX-Dx ICM system-related CFR at 30 days post-implant where the ICM system refers to the LUX-Dx ICM device, mobile applications, and the associated accessories used with the device. All implants and attempts with a de novo ICM are included in the at-risk group.
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | LUX-Dx PERFORM Study Enrollment
Number analyzed (Participants) | 687
Percentage of participants | 99.9 [99.0 to NA] — As prespecified in the study protocol the lower one-sided 97.5% confidence bound of the Kaplan-Meier estimate was compared to the performance goal (i.e., only the lower one-side confidence bound was necessary/utilized for hypothesis testing).

2. Primary Outcome: ICM System-related Complication-free Rate at 12 Months Post-implant
Time Frame: 12 months
Population: The chronic primary safety endpoint was the LUX-Dx ICM system-related CFR at 12 months post-implant where the ICM system refers to the LUX-Dx ICM device, mobile applications, and the associated accessories used with the device. All implants and attempts with a de novo ICM are included in the at-risk group.
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | LUX-Dx PERFORM Study Enrollment
Number analyzed (Participants) | 687
Percentage of participants | 99.6 [98.6 to NA] — As prespecified in the study protocol the lower one-sided 97.5% confidence bound of the Kaplan-Meier estimate was compared to the performance goal (i.e., only the lower one-side confidence bound was necessary/utilized for hypothesis testing).

ADVERSE EVENTS:
Time Frame: Adverse events were reported for all subjects following enrollment through their study end date. Subjects were considered to have completed the study after 12-Months of follow-up.
Arm/Group | LUX-Dx PERFORM Study Enrollment
All-Cause Mortality (participants affected / at risk) | 12/727
Serious Adverse Events (participants affected / at risk) | 127/727
Other Adverse Events (participants affected / at risk) | 152/727
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LUX-Dx PERFORM Study Enrollment (N=727)
1st Degree AV Block (Cardiac disorders) | 2 (2)
2nd Degree AV Block (Cardiac disorders) | 1 (1)
3rd Degree AV Block (Cardiac disorders) | 7 (7)
Abnormal Laboratory Values (General disorders) | 2 (2)
Atrial Fibrillation (AF) (Cardiac disorders) | 18 (26)
Atrial Flutter (Cardiac disorders) | 3 (4)
Atrial Tachycardia/Other SVT (e.g. AVRT, AVNRT, EAT) (Cardiac disorders) | 5 (5)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Cerebrovascular Accident (CVA) (Vascular disorders) | 9 (11)
Cerebrovascular accident (CVA) - ischemic (Vascular disorders) | 3 (3)
Chest Pain - Ischemic (Vascular disorders) | 2 (2)
Chest Pain - Other (General disorders) | 5 (7)
Coronary Artery Disease (Vascular disorders) | 2 (2)
Death (General disorders) | 2 (2)
Dehydration - Heart Failure (Cardiac disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema (Vascular disorders) | 1 (1)
Endocrine (Endocrine disorders) | 4 (7)
Fatigue/Weakness (General disorders) | 2 (2)
Fever and/or Virus (Infections and infestations) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 12 (14)
Genitourinary (Renal and urinary disorders) | 6 (6)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 3 (3)
Hematological (Blood and lymphatic system disorders) | 2 (2)
Hypertension/Hypertensive Crisis (Vascular disorders) | 1 (1)
Localized Infection (Infections and infestations) | 1 (2)
Multiple Heart Failure Symptoms (Cardiac disorders) | 9 (9)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 7 (7)
Myocardial Infarction (Vascular disorders) | 7 (7)
Neurological (Nervous system disorders) | 8 (9)
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 1 (1)
Pericardial effusion - unrelated procedure/device (Cardiac disorders) | 1 (1)
Physical Trauma (General disorders) | 2 (2)
Pleural Effusion - Heart Failure (Cardiac disorders) | 1 (3)
Pneumothorax - unrelated procedure/device (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Post Surgical wound discomfort/bruising/swelling (Injury, poisoning and procedural complications) | 1/718 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Renal (Renal and urinary disorders) | 8 (8)
Sinus Bradycardia (Cardiac disorders) | 9 (9)
Syncope (General disorders) | 8 (9)
System Infection (Infections and infestations) | 2 (2)
Transient Ischemic Attack (TIA) (Vascular disorders) | 4 (4)
Ventricular Fibrillation (VF) (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 1 (1)
Dislodgement - Unable to capture - RV (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LUX-Dx PERFORM Study Enrollment (N=727)
2nd Degree AV Block (Cardiac disorders) | 1 (1)
3rd Degree AV Block (Cardiac disorders) | 5 (5)
Adverse Reaction - other (Injury, poisoning and procedural complications) | 9/718 (9)
Atrial Fibrillation (AF) (Cardiac disorders) | 48 (50)
Atrial Flutter (Cardiac disorders) | 5 (5)
Atrial Tachycardia/Other SVT (e.g. AVRT, AVNRT, EAT) (Cardiac disorders) | 39 (72)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest Pain - Heart Failure (Cardiac disorders) | 1 (1)
Chest Pain - Other (General disorders) | 4 (6)
Coronary Artery Disease (Vascular disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea - Heart Failure (Cardiac disorders) | 2 (2)
Erosion (Product Issues) | 1/718 (1)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 1 (1)
Hypertension/Hypertensive Crisis (Vascular disorders) | 2 (2)
Hypotension/Orthostatic Hypotension (Vascular disorders) | 2 (2)
Infection (> 30 days post implant) (Infections and infestations) | 3/718 (3)
Integumentary (Skin and subcutaneous tissue disorders) | 2 (2)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Multiple Heart Failure Symptoms (Cardiac disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)
Neurological (Nervous system disorders) | 1 (1)
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 5 (5)
Other - ICM System (Product Issues) | 1/718 (1)
PG System - Patient Related - OTHER (Injury, poisoning and procedural complications) | 1/718 (1)
Patient Condition - Cardiovascular - OTHER (Cardiac disorders) | 1 (1)
Peripheral Vascular Disease (Vascular disorders) | 1 (2)
Post Surgical wound discomfort/bruising/swelling (Injury, poisoning and procedural complications) | 2/718 (2)
Post -Surgical infection ( 30 days post implant) (Injury, poisoning and procedural complications) | 4/718 (4)
Post-surgical pocket hemorrhage/bleeding/drainage (Injury, poisoning and procedural complications) | 4/718 (4)
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 26 (28)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 21 (21)
Syncope (General disorders) | 10 (13)
Transient Ischemic Attack (TIA) (Vascular disorders) | 3 (3)
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 3 (3)
Whole Body - OTHER (General disorders) | 2 (2)
Device Expulsion (Injury, poisoning and procedural complications) | 1/718 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT04732728/Prot_SAP_000.pdf